CLINICAL TRIAL: NCT06492863
Title: A Dose-escalation and Dose-expanded Phase I/II Clinical Study to Evaluate the Safety, and Efficacy of FT-003 in Subjects With Wet AMD
Brief Title: Gene Therapy(FT-003) for Wet AMD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Frontera Therapeutics (Industry)
Collaborators: Tianjin Medical University Eye Hospital (Other); The First Affiliated Hospital of Soochow University (Other); Peking Union Medical College Hospital (Other); Beijing Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FT003-C101
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: FT-003; nAMD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FT003 Dose 1 (Experimental): Low dose of FT-003
  Interventions: Genetic: FT-003
- FT003 Dose 2 (Experimental): Mid dose of FT-003
  Interventions: Genetic: FT-003
- FT003 Dose 3 (Experimental): High dose of FT-003
  Interventions: Genetic: FT-003

INTERVENTIONS:
Genetic: FT-003 — Administered via intraocular injection.

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability and efficacy of disposable vitreous injection of FT-003 in subjects with neovascular age-related Macular Degeneration (nAMD). The study was divided into two phases, Phase 1 dose escalation and Phase II dose expansion.

DETAILED DESCRIPTION:
FT-003 is a gene therapy product developed for the treatment of neovascular age-related macular degeneration (nAMD). Neovascular AMD is the main cause of blindness among elderly individuals. The available therapies for treating nAMD require life-long intravitreal (IVT) injections every 4-12 weeks to maintain efficacy. Administration of FT-003 has the potential to treat nAMD by providing durable expression of therapeutic levels of intraocular protein and maintaining the vision of patients. FT-003 is designed to reduce the current treatment burden which often results in undertreatment and vision loss in patients with nAMD receiving anti-VEGF therapy in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that are willing and able to follow study procedures;
* Female or male patients 50-80 years old at the time of signing the ICF;
* Clinically diagnosed with nAMD;
* Presence of active CNV
* The best corrected visual acuity (BCVA) of the studied eye is 24-73 letters;

Exclusion Criteria:

* •Presence of any other intraocular diseases other than nAMD in the studied eye that would affect the improvement of visual acuity and require treatment during the study for prevention or treatment of visual loss, as judged by the investigator.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2028-10-15 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability after FT-003 injection | At Week 12
  Incidence and severity of AE (Common Terminology Criteria for Adverse Events 5.0)

SECONDARY OUTCOMES:
To evaluate the efficacy after FT-003 injection | At Week 24
  the BCVA and OCT change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Xiaorong Li, Professor, Principal Investigator — Tianjin Medical University Eye Hospital
Locations (1):
- Tianjin Medical University Eye Hospital, Tianjin, Tianjin,China, China

IPD SHARING:
Plan to Share IPD: No